CLINICAL TRIAL: NCT03534401
Title: ARCHES Kenya: Addressing Reproductive Coercion in HEalth Settings
Brief Title: Addressing Reproductive Coercion in HEalth Settings - Kenya
Acronym: ARCHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); International Planned Parenthood Federation (Other); Population Council (Other)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor of Medicine and Global Public Health, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 170084
Record Dates: First submitted 2018-05-07; First posted 2018-05-23 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Unintended Pregnancy; Family Planning; Intimate Partner Violence (IPV)
Keywords: Reproductive Coercion; Gender-based violence; Contraception; Clinic-based screening for IPV; Clinic-based counseling

STUDY DESIGN:
Intervention Model Description: The ARCHES Kenya study will take place in six IPPF-affiliated Family Health Options Kenya (FHOK) clinics in Nairobi, Kenya or surrounding smaller cities for all clients receiving voluntary FP counseling. The intervention study will involve a matched cluster control trial. Three clinics will serve as the intervention sites and three other clinics matched on client volume and demographics, clinic structure and staffing will serve as matched comparison sites and will not receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Contraceptive Counseling (No Intervention): Providers at control clinics receive no additional training; clients receive standard contraceptive counseling services.
- ARCHES Kenya Intervention in Contraceptive Counseling (Experimental): Providers at intervention clinics receive training on ARCHES strategies integrated into contraceptive counseling; clients receive the ARCHES Kenya intervention integrated within standard contraceptive counseling services.
  Interventions: Behavioral: ARCHES Kenya

INTERVENTIONS:
Behavioral: ARCHES Kenya — ARCHES: Contraceptive counselors in intervention clinics will receiving training to ) provide counseling and education regarding risk of partner detection of contraceptive methods, and women's and girls' strategies to use contraceptive methods to minimize partner detection risk integrated into standard contraceptive counseling, b) make brief inquiries to allow clients the opportunity to disclose experiences of RC and IPV (i.e., screening), c) provide method-specific counseling based on this information and the method chosen by the client, d) provide supported linkage of IPV survivors to local IPV support services (i.e. warm referral), and e) offer palm-sized educational materials on RC and IPV, as well as IPV services to all clients.
  Arms: ARCHES Kenya Intervention in Contraceptive Counseling

SUMMARY:
The primary purpose of this research is to conduct a small matched cluster control trial of an intervention designed to address reproductive coercion and unintended pregnancy (ARCHES - Addressing Reproductive Coercion within Healthcare Settings) adapted to the Kenyan cultural and family planning healthcare context (ARCHES Kenya) so as to provide initial data regarding acceptability, feasibility and efficacy in this high-need LMIC context.

DETAILED DESCRIPTION:
The project consortium will implement the ARCHES Kenya model across 6 Family Health Options Kenya clinics in Nairobi, Kenya. A matched-pair cluster control design including 600 female family planning (FP) clients ages 15-49 years (inclusive of 360 clients age 15-24 years) will be utilized to evaluate this intervention. Baseline data will be collected prior to routine FP service delivery, with a short exit survey conducted immediately following the clients' FP appointment (ARCHES or standard FP counseling will be provided during this visit). Follow-up data will be collected at 3 and 6-months post-intervention. Qualitative data will be collected from intervention providers (n=12) regarding implementation via weekly technical assistance sessions during the first three months, and then monthly, regarding acceptability and feasibility of integrating ARCHES into routine FP counseling, including barriers and facilitators to implementation, and any issues with maintaining fidelity to the ARCHES model. Structured interviews with select providers (n=12) will also be conducted at 3-months post-training to delve further into these issues. Structured interviews with intervention participants reporting experience of RC in the past 3 months on the baseline survey (20 participants ages 15-24, 15 ages 25-49; total n=35) will be conducted at 3-months follow-up to assess their experience of the intervention; perceived utility of the messages, care and materials; barriers to utilizing messaging and materials; and suggestions for improvement. Analyses specific to participants ages 15-24 will provide findings to guide consideration of ARCHES as an effective strategy to improve reproductive health and reduce GBV among adolescents in the region. The project consortium will engage Government of Kenya officials, IPPF executive directors and IPPF member associations across the federation to pave the way for the future roll out of this approach in other low and middle-income country (LMIC) contexts.

ELIGIBILITY:
Inclusion Criteria:

* Visiting FHOK study clinic "for family planning or interested in receiving family planning"
* Aged 15-49 years
* Not currently pregnant (self-report)
* Not sterilized (self-report)
* Have a male partner with whom they have had sex in the past 3 months
* Biologically Female
* Not planning to move out of the area in the next 6 months
* Have a mobile phone that can be safely used for recontacting
* Able to safely participate in a private interview

Exclusion Criteria:

* Declined to participate
* Participated in pilot (measured by taking a women's health survey at the clinic in the past 3 months)
* Unable or unwilling to complete exit survey, or reported not receiving any contraceptive counseling at exit

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — self-report biologically female
Enrollment: 659 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Reproductive Coercion | Change from baseline number reporting reproductive coercion at 3 and 6 month follow-up (combined)
  Binary (yes/no) measure based on 9-item indicator list (entitled the Reproductive Coercion Scale) assessing incidence of male partner behaviors that interfere with or prevent use of contraception or coerce pregnancy in prior 3 months. A "yes" response to any of the 9-items indicates reproductive coercion is present.
Number of Participants Reporting Intimate Partner Violence | Change from baseline number reporting physical intimate partner violence at 3 and 6 month follow-up (combined)
  Binary (yes/no) measure based on adapted version of the injury subscale of the Conflict Tactics Scale 2 (CTS-2). A "yes" response to any of the subscale items indicates physical intimate partner violence is present.
Number of Participants Reporting Sexual Intimate Partner Violence | Change from baseline number reporting sexual intimate partner violence at 3 and 6 month follow-up (combined)
  Binary (yes/no) measure based on single item modified from the Sexual Experiences Short-Form Survey. A "yes" response to this item indicates sexual intimate partner violence is present.
Number of Participants Reporting Uptake of a Modern Contraceptive Method | Assessed at exit interview on month 0 (immediately after baseline and provider appointment)
  Binary (yes/no) measure based on response if participant received a method from their provider and reported a modern method (IUD, implant, injection, pill, condom). A "yes" response to receiving a method and receiving one of the modern methods listed indicates update a modern contraceptive method.

SECONDARY OUTCOMES:
Number of Participants Reporting Incident Pregnancy | Assessed at 3 months and 6 month follow-up (combined)
  Binary (yes/no) measure based on one self-report item asking how many times client has been pregnant in past 3 months. A response of greater than zero indicates incident pregnancy.
Number of Participants Reporting Incident Unintended Pregnancy | Assessed at 3 months and 6 month follow-up (combined)
  Binary (yes/no) measure based on an additional item for those self-reporting incident pregnancy "at the time you became pregnant, did you want to become pregnant then, did you want to wait to become pregnant at a later date, or did you not want any more children?" A response of "wanted to wait until later date" OR "did not want anymore children" for incident pregnancy in prior 3 months indicates incident unintended pregnancy.
Mean Contraception Self-efficacy Including in the Face of Reproductive Coercion Scale Score (1) | Change from baseline mean contraceptive self-efficacy score at 3 month follow-up
  Investigator developed contraceptive self-efficacy scale, 4-items, Likert response (strongly agree, somewhat agree, disagree), sum score minimum 0 to maximum 8. Higher score indicates better outcome (i.e., greater contraceptive self-efficacy).
Mean Contraception Self-efficacy Including in the Face of Reproductive Coercion Scale Score (2) | Change from baseline mean contraceptive self-efficacy score at 6 month follow-up
  Investigator developed contraceptive self-efficacy scale, 4-items, Likert response (strongly agree, somewhat agree, disagree), sum score minimum 0 to maximum 8. Higher score indicates better outcome (i.e., greater contraceptive self-efficacy).
Mean Attitudes Justifying Reproductive Coercion Scale Score (1) | Change from baseline mean attitudes justifying reproductive coercion score at 3 month follow-up
  Investigator developed scale measuring attitudes justifying reproductive coercion. Sum score based on 8-item scale (minimum 0, maximum 8) asking participants if it is acceptable for husbands or male partners to enact different forms of RC in a variety of situations, based on participant response to agree/disagree and summed number of agrees over the items. Higher scores indicate worse outcome (i.e., greater justification of reproductive coercion).
Mean Attitudes Justifying Reproductive Coercion Scale Score (2) | Change from baseline mean attitudes justifying reproductive coercion score at 6 month follow-up
  Investigator developed scale measuring attitudes justifying reproductive coercion. Sum score based on 8-item scale (minimum 0, maximum 8) asking participants if it is acceptable for husbands or male partners to enact different forms of RC in a variety of situations, based on participant response to agree/disagree and summed number of agrees over the items. Higher scores indicate worse outcome (i.e., greater justification of reproductive coercion).
Mean Attitudes Justifying Intimate Partner Violence Scale Score (1) | Change from baseline mean attitudes justifying intimate partner violence score at 3 month follow-up
  Adapted scale measuring attitudes justifying intimate partner violence. Sum score (minimum 0, maximum 7) based on adapted DHS justification of wife beating scale (7-items), based on participant response to agree/disagree and summed number of agrees over the items. Higher scores indicate worse outcome (i.e., greater justification of intimate partner violence).
Mean Attitudes Justifying Intimate Partner Violence Scale Score (2) | Change from baseline mean attitudes justifying intimate partner violence score at 6 month follow-up
  Adapted scale measuring attitudes justifying intimate partner violence. Sum score (minimum 0, maximum 7) based on adapted DHS justification of wife beating scale (7-items), based on participant response to agree/disagree and summed number of agrees over the items. Higher scores indicate worse outcome (i.e., greater justification of intimate partner violence).
Number of Participants Reporting Awareness of Intimate Partner Violence Services (1) | Change from baseline number reporting awareness of intimate partner violence services at 3 month follow-up
  Binary (yes/no) measure based on four-items assessing reported awareness of listed local services for women and girls experiencing IPV. A "yes" response to any of the four items indicates awareness of IPV services.
Number of Participants Reporting Awareness of Intimate Partner Violence Services (2) | Change from baseline number reporting awareness of intimate partner violence services at 6 month follow-up
  Binary (yes/no) measure based on four-items assessing reported awareness of listed local services for women and girls experiencing IPV. A "yes" response to any of the four items indicates awareness of IPV services.
Number of Participants Reporting Covert Use of Contraceptives (1) | Change from baseline number reporting covert use of contraceptives at 3 month follow-up
  Binary (yes/no) measure based on one item if a client has "used family planning without telling a male partner" in the past 3 months. A "yes" response indicates covert use of contraceptives in the past 3 months. Assessed for all clients and those reporting RC/IPV separately.
Number of Participants Reporting Covert Use of Contraceptives (2) | Change from baseline number reporting covert use of contraceptives at 6 month follow-up
  Binary (yes/no) measure based on one item if a client has "used family planning without telling a male partner" in the past 3 months. A "yes" response indicates covert use of contraceptives in the past 3 months. Assessed for all clients and those reporting RC/IPV separately.
Utilization of Intimate Partner Violence Services | Assessed at 3 months and 6 month follow-up (combined)
  Binary (yes/no) measure based on items assessing whether a participant called or visited a listed local service for women or girls experiencing IPV in the past 3 months. A "yes" response indicates utilization of IPV services in the past 3 months. Assessed for all clients and those reporting RC/IPV separately.
Leaving a Relationship Because it Felt Unsafe, Unhealthy or Abusive | Assessed at 3 months and 6 month follow-up (combined)
  Binary (yes/no) measure based on question "in the last three months, have you left a relationship because it felt unhealthy, unsafe, or abusive?" A "yes" response indicates leaving a relationship because it felt unsafe, unhealthy, or abusive. Assessed for all clients and those reporting RC/IPV separately.

CONTACTS AND LOCATIONS:
Overall Officials: Jay G Silverman, PhD, Principal Investigator — UCSD Center on Gender Equity and Health
Locations (1):
- Center on Gender Equity and Health, University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data included in analyses will be shared in a public data repository at the time of publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The study protocol was published in 2020 prior to completion of data collection (https://doi.org/10.1186/s12978-020-00916-9). Informed consent forms and analytic code will be made available at the time of publication.

REFERENCES:
- [Derived] Uysal J, Schwarz E, Liambila W, Wendoh S, Fonseka RW, Monroy RV, Boyce SC, Pearson E, Silverman JG. Strategies to address reproductive coercion and intimate partner violence in Nairobi family planning services: qualitative client and provider perspectives. Sex Reprod Health Matters. 2025 Dec;33(1):2570528. doi: 10.1080/26410397.2025.2570528. Epub 2025 Dec 15. PMID 41070626
- [Derived] Uysal J, Carter N, Johns N, Boyce S, Liambila W, Undie CC, Muketo E, Adhiambo J, Gray K, Wendoh S, Silverman JG. Protocol for a matched-pair cluster control trial of ARCHES (Addressing Reproductive Coercion in Health Settings) among women and girls seeking contraceptive services from community-based clinics in Nairobi, Kenya. Reprod Health. 2020 May 27;17(1):77. doi: 10.1186/s12978-020-00916-9. PMID 32460786